CLINICAL TRIAL: NCT05601388
Title: Role of IMP3 Expression in Colorectal Carcinoma: An Immunohistochemical Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagwa Abd El-Sadek Ahmed, Lecturer at Pathology Department, Faculty of Medicine, Sohag University
Other Study IDs: Soh-Med-22-09-16
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months

SUMMARY:
Colorectal carcinoma (CRC) is the third most common malignancy worldwide. In Egypt, the relative frequency of CRC is about 9-12% with high male predominance 3:1. The high mortality rates associated with CRC is reflective of several factors including: the lack of apparent symptoms in the early stages and the absence of cancer prevention strategies in developing countries.

Insulin-like growth factor II m-RNA-binding protein 3 (IMP3) is a member of the IMP family which plays a key role in the transfer and stabilization of mRNA, cell growth, and migration during embryogenesis. IMP3 has gained considerable interest as a cancer-associated protein. Previous studies strongly suggest that IMP3 may represent a valuable prognostic marker in human cancer. Its overexpression has been reported in a variety of human types of cancer, including lung cancer, colon cancer, pancreatic cancer, gastric cancer, liver cancer, and breast cancer

DETAILED DESCRIPTION:
Colorectal carcinoma (CRC) is the third most common malignancy worldwide. In Egypt, the relative frequency of CRC is about 9-12% with high male predominance 3:1. The high mortality rates associated with CRC is reflective of several factors including: the lack of apparent symptoms in the early stages and the absence of cancer prevention strategies in developing countries.

Insulin-like growth factor II m-RNA-binding protein 3 (IMP3) is a member of the IMP family which plays a key role in the transfer and stabilization of mRNA, cell growth, and migration during embryogenesis. To date, there are three known members of IMP family proteins: IMP1, IMP2, and IMP3 . IMP3 has gained considerable interest as a cancer-associated protein. Previous studies strongly suggest that IMP3 may represent a valuable prognostic marker in human cancer. Its overexpression has been reported in a variety of human types of cancer, including lung cancer, colon cancer, pancreatic cancer, gastric cancer, liver cancer, and breast cancer

It has been reported that IMP3 expression, determined via immunohistochemistry (IHC), has prognostic significance in CRC, recent studies revealed that IMP3 expression in tumor cells is a marker of poor prognosis in CRC patients and promotes tumor cell proliferation, adhesion, and invasion. Despite these observations, the IMP3 expression and its clinicopathologic significance in human CRC needs further elucidation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CRC and will be underwent surgery.

Exclusion Criteria:

* - Patients received pre-operative chemotherapy or radiotherapy.
* Patients with insufficient clinical data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Sixty specimens of CRC will be obtained from patients who will undergo colectomy in General Surgery Department of Sohag Faculty of Medicine according to local Ethical Committee regulations, to be examined in the Pathology Laboratory of the same faculty. From October 2022, till completing the sample size.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
evaluate the immunohistochemical (IHC) expression of IMP3 in CRC and to correlate its expression with some known clinicopathological parameters. | 4 months
  IHC

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag, Egypt